CLINICAL TRIAL: NCT05754905
Title: High-resolution Contrast-enhanced Magnetic Mesonance Angiography of Children's Hip Joint
Brief Title: High-resolution CE-MRA of Children's Hip Joint
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuxi Su, Orthopaedic Department, Children's Hospital of Chongqing Medical University
Other Study IDs: CQMU-2023-2
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Hip; Vessels; Anomaly; Magnetic Resonance; Three-dimensional Water-selective Cartilage (3D-WATSc)
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal hip joint: The normal side of patients with hip joint disease
  Interventions: Other: Magnetic resonance examination
- Abnormal hip joint: The abnormal side of patients with hip joint disease
  Interventions: Other: Magnetic resonance examination

INTERVENTIONS:
Other: Magnetic resonance examination — the two groups are underwent magnetic resonance examination including enhanced 3D-WATSc sequence

SUMMARY:
The goal of this observational study is to learn about the feasibility of enhanced three-dimensional water-selective cartilage (3D-WATSc) sequence in displaying the vessels of children's hip by magnetic resonance. The main questions it aims to answer are:

* Could the images of enhanced 3D-WATSc sequence show the healthy side hip joint vessels in children?
* Could the images of enhanced 3D-WATSc sequence show the vascular disease of the suffering side hip joint in children?

Participants with unilateral hip disease will undergo the magnetic resonance examination including enhanced 3D-WATSc sequence. The pelvic plain film and magnetic resonance images will be collected and analysed.

Researchers will compare the images of of the normal side with the images of the abnormal side to see if the enhanced 3D-WATSc sequence images could show the vascular disease of the suffering side hip joint in children?

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months-14 years who are diagnosed as hip disease after screening by pediatric orthopedic surgeon in Children's Hospital of Chongqing Medical University during the study period. The hip disease contain developmental dysplasia of the hip, Perthes disease, infection of the hip, inflammation of the hip, fracture of the hip, and Meyer's dysplasia.

Exclusion Criteria:

* patients with bilateral hip joint disease; patients with claustrophobia;Patients with metal implants (such as pacemaker implantation)

Ages: 6 Months to 14 Years | Sex: All
Age Groups: Child
Study Population: Children with hip disease from 2021-2022 in Children's Hospital of Chongqing Medical University
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
The medial circumflex femoral artery (MCFA) and lateral circumflex femoral artery (LCFA) of the bilateral hip joint | 1 day (Magnetic resonance examination end time)
  Morphology of the MCFA and LCFA of the bilateral hip joint
The branches of the MCFA and/or LCFA around the bilateral femoral neck | 1 day (Magnetic resonance examination end time)
  Morphology of MCFA and/or LCFA branches around the bilateral femoral neck
The vessels of secondary ossification center and/or cartilaginous vascular canal in bilateral femoral head | 1 day (Magnetic resonance examination end time)
  Morphology of the vessels and cartilaginous vascular canal in bilateral femoral head

CONTACTS AND LOCATIONS:
Overall Officials: Yuxi Su, M.D., Study Chair — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No